CLINICAL TRIAL: NCT02754635
Title: Induction of Labor at Term Versus Expectant Management Among Women With Abnormal Maternal Serum Biochemical Markers: A Randomized Controlled Trial
Brief Title: Induction Versus Expectant Management With Abnormal Maternal Biochemical Markers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Manal Massalha, Principal Investigator, HaEmek Medical Center, Israel
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 00126-15-EMC
Record Dates: First submitted 2016-02-23; First posted 2016-04-28 (Estimated); Last update posted 2017-08-16 (Actual); Status verified 2017-08

CONDITIONS: PREGNANCY
Keywords: Abnormal first or second trimester biochemical markers; maternal and perinatal morbidity/mortality
MeSH Terms: interventions — Labor, Induced; Watchful Waiting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Induction of labour (Active Comparator): Induction of labour at 38-39 weeks
  Interventions: Other: Induction of labour
- Expectant management (Active Comparator): Expectant management until 41 weeks.
  Interventions: Other: Expectant management

INTERVENTIONS:
Other: Induction of labour — Induction of labour
  Arms: Induction of labour
Other: Expectant management — Expectant management
  Arms: Expectant management

SUMMARY:
Induction of labor at term versus expectant management among women with abnormal maternal biochemical markers. A randomized controlled trial

DETAILED DESCRIPTION:
Pregnancy-associated plasma protein A (PAPP-A), alpha-fetoprotein (AFP), human chorionic gonadotropin (hCG), and inhibin A, are biochemical markers that are part of the first and second trimester screening test, for Down syndrome and neural tube defects in pregnancy. These biochemical markers have been shown also to be associated with slightly increased risk for adverse pregnancy outcomes in the absence of aneuploidy or neural tube defects, for example; preeclampsia, low birth weight, placental abruption, preterm labor, and intrauterine fetal death.

There are no guidelines regarding the management of these cases assuming a reassuring maternal and fetal status are normal, at term (38 - 39 weeks). However, adverse events may still develop between 38 to 42 weeks when calculated according to ongoing pregnancy.

Investigators aim in this randomized trial to examine the effect of induction of labor at 38 - 39 weeks compared to expectant management among women with abnormal first or second biochemical screening tests on maternal and perinatal outcomes.

Enrollment: 320 women in both groups. Interim analyses will be performed after enrolling 50% of the participants.

ELIGIBILITY:
Inclusion Criteria:

* HCG, AFP or Inhibin greater than 2 multiple of median (MOM) or PAPPA less than 0.15 MOM.
* Singleton.
* Appropriate for gestational age fetus.
* Reassuring fetal status including normal amniotic fluid index.

Exclusion Criteria:

* Any hypertensive disorder.
* Indication for induction of labour at enrollment.
* Any contraindication of induction of labour.
* Prior cesarean delivery.
* Any contraindication for a trial of vaginal delivery.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 320 (Estimated)
Dates: Start 2016-03; Primary Completion 2018-05 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Placental abruption | 4 weeks
  Clinical diagnosis. Co-primary endpoint #1.
Gestational hypertension | 4 weeks
  Blood pressure above 140/90 mmHg. Co-primary endpoint #2
Small of gestational age | 4 weeks
  Birth Weight less than the 10th percentile. Co-primary endpoint #3
Intra-uterine death | 4 weeks
  Fetal death. Co-primary endpoint #4

SECONDARY OUTCOMES:
Mode of delivery | 4 weeks
  vaginal or cesarean.
Intrapartum fever | 4 weeks
  fever above 38C
Neonatal Apgar score | 4 weeks
  Apgar score

CONTACTS AND LOCATIONS:
Overall Officials: Raed Salim, Study Chair — Emek Medical Center
Locations (1):
- Emek medical center, Afula, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Yuan W, Chen L, Bernal AL. Is elevated maternal serum alpha-fetoprotein in the second trimester of pregnancy associated with increased preterm birth risk? A systematic review and meta-analysis. Eur J Obstet Gynecol Reprod Biol. 2009 Jul;145(1):57-64. doi: 10.1016/j.ejogrb.2009.04.017. Epub 2009 May 19. PMID 19457604
- [Result] Ganapathy R, Lamont RF, Bassett P. Unexplained elevated maternal serum beta-HCG concentration and adverse pregnancy outcome. Prenat Diagn. 2007 Nov;27(11):995-9. doi: 10.1002/pd.1813. PMID 17621365
- [Result] Alkazaleh F, Chaddha V, Viero S, Malik A, Anastasiades C, Sroka H, Chitayat D, Toi A, Windrim RC, Kingdom JC. Second-trimester prediction of severe placental complications in women with combined elevations in alpha-fetoprotein and human chorionic gonadotrophin. Am J Obstet Gynecol. 2006 Mar;194(3):821-7. doi: 10.1016/j.ajog.2005.09.010. PMID 16522419
- [Result] Gagnon A, Wilson RD; SOCIETY OF OBSTETRICIANS AND GYNAECOLOGISTS OF CANADA GENETICS COMMITTEE. Obstetrical complications associated with abnormal maternal serum markers analytes. J Obstet Gynaecol Can. 2008 Oct;30(10):918-932. doi: 10.1016/S1701-2163(16)32973-5. English, French. PMID 19038077
- [Result] Luckas MJ, Sandland R, Hawe J, Neilson JP, McFadyen IR, Meekins JW. Fetal growth retardation and second trimester maternal serum human chorionic gonadotrophin levels. Placenta. 1998 Mar-Apr;19(2-3):143-7. doi: 10.1016/s0143-4004(98)90002-9. PMID 9548180
- [Result] Wax JR, Lopes AM, Benn PA, Lerer T, Steinfeld JD, Ingardia CJ. Unexplained elevated midtrimester maternal serum levels of alpha fetoprotein, human chorionic gonadotropin, or low unconjugated estriol: recurrence risk and association with adverse perinatal outcome. J Matern Fetal Med. 2000 May-Jun;9(3):161-4. doi: 10.1002/1520-6661(200005/06)9:33.0.CO;2-T. PMID 10914623
- [Result] Salim R, Okopnik M, Garmi G, Nachum Z, Zafran N, Shalev E. Lack of association between unexplained elevated maternal serum alpha fetoprotein and/or human chorionic gonadotropin and the occurrence of placental thrombotic lesions. Placenta. 2010 Apr;31(4):277-81. doi: 10.1016/j.placenta.2010.01.010. Epub 2010 Feb 4. PMID 20132984
- [Result] Saruhan Z, Ozekinci M, Simsek M, Mendilcioglu I. Association of first trimester low PAPP-A levels with adverse pregnancy outcomes. Clin Exp Obstet Gynecol. 2012;39(2):225-8. PMID 22905470
- [Result] Dugoff L, Hobbins JC, Malone FD, Vidaver J, Sullivan L, Canick JA, Lambert-Messerlian GM, Porter TF, Luthy DA, Comstock CH, Saade G, Eddleman K, Merkatz IR, Craigo SD, Timor-Tritsch IE, Carr SR, Wolfe HM, D'Alton ME; FASTER Trial Research Consortium. Quad screen as a predictor of adverse pregnancy outcome. Obstet Gynecol. 2005 Aug;106(2):260-7. doi: 10.1097/01.AOG.0000172419.37410.eb. PMID 16055573
- [Result] Caughey AB, Stotland NE, Escobar GJ. What is the best measure of maternal complications of term pregnancy: ongoing pregnancies or pregnancies delivered? Am J Obstet Gynecol. 2003 Oct;189(4):1047-52. doi: 10.1067/s0002-9378(03)00897-4. PMID 14586353
- [Result] Hossain N, Paidas MJ. Adverse pregnancy outcome, the uteroplacental interface, and preventive strategies. Semin Perinatol. 2007 Aug;31(4):208-12. doi: 10.1053/j.semperi.2007.05.002. PMID 17825674
- [Result] Konchak PS, Bernstein IM, Capeless EL. Uterine artery Doppler velocimetry in the detection of adverse obstetric outcomes in women with unexplained elevated maternal serum alpha-fetoprotein levels. Am J Obstet Gynecol. 1995 Oct;173(4):1115-9. doi: 10.1016/0002-9378(95)91336-x. PMID 7485303